CLINICAL TRIAL: NCT05057156
Title: Digital Solution to Improve Cognitive Function in Epilepsy: PRODDIGE Project
Acronym: PRODDIGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020PI095; 2020-A02482-37 (Registry Identifier: ID RCB)
Record Dates: First submitted 2021-06-29; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-05

CONDITIONS: Cognitive Change
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: multicentric, transversal and randomized trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "application supervised by a psychologist via teleconsultations" (Experimental): patient have app, and teleconsultation with psychologist
  Interventions: Behavioral: cognitive rehabilitation
- "application in total autonomy" (Placebo Comparator): patients have app, they play when they want
  Interventions: Behavioral: cognitive rehabilitation
- "control" group without using the application (No Intervention): patients haven't app

INTERVENTIONS:
Behavioral: cognitive rehabilitation — patients have to use an app with cognitive games
  Arms: "application in total autonomy"; "application supervised by a psychologist via teleconsultations"

SUMMARY:
Background: Epilepsy leads to cognitive impairment in 20-50%. Compared to seizures, these cognitive disorders are a major additional factor in occupational, social and family disability. Memory and language skills are most often impaired. These disorders are well described, multifactorial, but no therapy (drug and/or non-drug) has been validated to date. Recently, cognitive remediation techniques have shown benefits in certain neurological pathologies, such as multiple sclerosis. In adult epilepsy, few previous cognitive remediation studies were performed but suffer significant methodological shortcomings that limit the scope of their results. Studies that have focused on cognitive function have shown promising results for attention and memory. In contrast, in the area of language, no studies have been published.

Objective: to evaluate the effectiveness of a digital solution (PRODDIGE*) on the lexical access capacities in people with epilepsy.

Method: Randomized, multicentric, observational study which will compare the use of a digital solution (PRODDIGE) in total autonomy versus the supervised use by a trained neuropsychologist. A neuropsychological assessment will be provided before and after a period of 4 months of use of the digital solution.

Material: The medical project aims to offer an application of cognitive remediation to patients who suffer from cognitive impairments and especially language disorders.

T The App is like a serious game, it's based on the playfulness of "game" and the seriousness of "medical exercise". During the exercise the patient can ask for clues help and isn't constrained by time in order to succeed "his mission".

Conclusion: This will be the first French speaking app specifically dedicated to rehabilitation of language deficits observed in people with epilepsy. The expected benefits are an improvement of the patients' language complaints, the regular use of an adapted digital solution to improve their language difficulties, but also a better understanding of their disorders and an improvement of their self-esteem.

DETAILED DESCRIPTION:
o best help patients, Norsys enterprise designed the app with three key principles:

1. Co-designed, to encourage the emergence of original solutions about uses from patients and therapists,
2. User-friendly, to encourage the patient to exercise regularly and with pleasure (soft, optimistic, pleasant and calm mood),
3. Accessible design, to get an application compatible and adapted to the specifics of these patients (contrast, color, typography, manipulation) According to these principles, the app gives access to 6 mini-games in its first version and will be available on iOS and Android smartphones.

These exercises allow patients to work on specific aspects of their pathologies, this is how the exercises are intended to be playful, dynamic (ex. drag'n'drop) and sometimes collaborative.

ELIGIBILITY:
Inclusion Criteria:

* Person with epilepsy, according to Fisher et al. (2005) criteria: all type of epilepsy could be include (new-onset and drug-resistant)
* Treatment must have been stable for 4 months: have the same molecule
* Person who has received full information about the organization of the research and has not objected to his or her participation and the use of his or her data
* Person aged 18 and over
* Mandatory affiliation to a social security scheme
* Validated cognitive inclusion criterion: having a YES response on the cognitive complaint questionnaire :

A.Spontaneous complaint :

Does the patient spontaneously complain of language difficulties?

B.Subjective complaint :

1. Do you search for your words?
2. Do you sometimes feel like you have the word on the tip of your tongue?
3. Do you sometimes have trouble finding the names of people you know well?
4. Do you ever say one word for another?

Exclusion Criteria:

* Person with another neurological condition

Patients and normal control :

* A person over the age of majority who is subject to a legal protection measure or who is unable to express their consent.
* Person deprived of liberty by a judicial or administrative decision
* A person who regularly uses psychoactive substances (cannabis, alcohol, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Number of weekly connections of epileptic patients in each group. | 5 months
  Evaluate the compliance to the digital application by counting the number of connections

SECONDARY OUTCOMES:
Feeling the frequency of lexical access problems | 0 and 5 months
  Interview : Questionnaire language score : 0 to 12 points : 12 = worse outcome
Self-esteem assessment | 0 and 5 months
  Interview : Self-esteem score (Rosenberg scale) 0 to 40 points : 40 = better outcome
Mood assessment | 0 and 5 months
  Depression scale score (Neurological Disorder Depression Inventory for Epilepsy : NDDI-E) : 6 to 24 points : 24 = worse outcome
Anxiety assessment | 0 and 5 months
  Anxiety scale score : (Generalized Anxiety Disorder: GAD-7) : 0 to 21 points : 21 = worse outcome
Information processing speed | 0 and 5 months
  Computerized Speed Cognitive Test (CSCT): processing speed index: number of correct items in 90 sec. 0 to 110 points : 110 = better outcome
Lexicon access assessment | 0 and 5 months
  Lexicon access tests (Denomination Orale 80): number of correctly named words (0 to 80 words) : 80 = better outcome
lexicon access assessment in time | 0 and 5 months
  Lexicon access tests (Denomination Orale 80): time in second
Selective and sustained attention assessment | 0 and 5 months
  Selective Attention Test: Paced Auditory Serial Audition Test 4 seconds (PASAT): 0 to 60 score : 60 = better outcome
Working memory assessment | 0 and 5 months
  Backward digit span: number of digits recalled correctly in inverse order: 0 to 9 score: 9 = better outcome
Verbal fluency assessment | 0 and 5 months
  Verbal Initiation Test: Phonological Fluency: number of words beginning with P given in 2 minutes 0 to 50 words Category fluency test: number of words given in 2 minutes that belong to the category of Animals.0 to 50 words
Naming assessment Boston naming task | 0 and 5 months
  Number of correctly named words Boston Naming Test: number of correctly named words :0 to 50 points : 50 = better outcome
Naming assessment in time | 0 and 5 months
  Number of correctly named words Boston Naming Test: time in second
Naming assessment BETL | 0 and 5 months
  Number of correctly named words (BETL task : batterie evaluation troubles lexicaux = assessment of lexical impairment battery) 0 to 54 point : 54 = better outcome
Naming assessment BETL intime | 0 and 5 months
  BETL task : batterie evaluation troubles lexicaux = assessment of lexical impairment battery) : time in second

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT05057156/Prot_000.pdf